CLINICAL TRIAL: NCT05133505
Title: Characterisation of TIM-3/Gal-9 Immune Checkpoints in Primary Central Nervous System Diffuse Large B Cell Lymphomas
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0665
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary central nervous system diffuse large B cell lymphoma is a rare and aggressive entity of diffuse large B cell lymphoma. A previous transcriptomic study showed an overexpression of TIM-3 and Gal-9 in the tumor microenvironment. The investigators aimed to characterise TIM-3/Gal-9 immune checkpoints by using immunohistochemistry in the tumor microenvironment of primary central nervous system diffuse large B cell lymphoma.

ELIGIBILITY:
Inclusion criteria:

- patient with a Diagnosis of LBDGC-SNC

Exclusion criteria:

* immunocompromised patients
* patients with a history of previous or associated low-grade lymphoma
* patients with a history of systemic LBDGC with secondary localization to the SNC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient of Primary central nervous system diffuse large B cell lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
TIM-3 and Gal-9 immunohistochemical expression | 1 day
  TIM-3 and Gal-9 immunohistochemical expression by tumor and microenvironment cells

CONTACTS AND LOCATIONS:
Overall Officials: aline desrumaux, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC